CLINICAL TRIAL: NCT01291550
Title: Electronic Nose for Diagnosis of Neurodegenerative Diseases Via Breath Samples
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Prof Judith aharon-Peretz, Rambam Medica Center
Other Study IDs: 0196-09
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2010-09

CONDITIONS: Neurodegenerative Diseases
Keywords: Detecting volatile biomarkers using breath sample
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Nerodegenerative diseases: Patients with parkinsonism and patients with dementia
- Controls
- ADHD: Subjects diagnosed with ADHD

SUMMARY:
The diagnosis of neurodegenerative conditions and ADHD still mostly relies on clinical symptoms as there are no validated, inexpensive, and simple bio- markers available yet. The purpose of this study is to deliver a proof-of-concept for novel biomarkers to identify neurodegenerative conditions and ADHD based on breath testing.

Alveolar breath will be collected from healthy volunteers, patients with extrapyramidal conditions, patients diagnosed with dementia and from ADHD subjects. The discriminative power of a tailor-made Nanoscale Artificial Nose (™NA-NOSE) containing an array of six nanomaterial-based sensors will be tested. Discriminant factor analysis will be applied to the NA-NOSE signals in order to detect statistically significant differences between the sub-populations, and classification success will be estimated using leave-one-out cross-validation. The identification of NA-NOSE patterns will be supported by analyzing the chemical composition of the breath using gas-chromatography in conjunction with mass-spectrometry (GC-MS).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with neurodegenerative conditions
* Healthy subjects
* Subjects diagnosed with ADHD

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Out patient clinic patients diagnosed with neurodegenerative conditions healthy control and subjects diagnosed with ADHD.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-09

CONTACTS AND LOCATIONS:
Locations (1):
- Cognitive Neurology, Rambam Medical Center, Haifa, Israel

REFERENCES:
- [Derived] Tisch U, Schlesinger I, Ionescu R, Nassar M, Axelrod N, Robertman D, Tessler Y, Azar F, Marmur A, Aharon-Peretz J, Haick H. Detection of Alzheimer's and Parkinson's disease from exhaled breath using nanomaterial-based sensors. Nanomedicine (Lond). 2013 Jan;8(1):43-56. doi: 10.2217/nnm.12.105. Epub 2012 Oct 15. PMID 23067372